CLINICAL TRIAL: NCT05144776
Title: Evaluation of Novel Hepatitis B DNA Test from Capillary Blood At the Point-of-care As a Tool to Enhance Clinical Management
Brief Title: Evaluation of Hepatitis B Virus (HBV) DNA Test As Point of Care Tool
Acronym: HBVPOCT
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Responsible Party: Sponsor
Other Study IDs: VHCRP 2103
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Dried blood spot samples will collected, tested for HBV viral load and remaining samples stored for future unspecified ethically approved HBV research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic hepatitis B: 300 patients diagnosed with chronic hepatitis B will be enrolled. A fingerstick HBV DNA test will be performed using the Xpert HBV Viral Load assay, and a dried blood spot sample will be collected which will be tested using a gold standard HBV DNA viral load assay. Both results will be compared against the HBV DNA viral load from standard of care venous blood using the gold standard HBV DNA viral load assy. Enrolment of HBV DNA undetectable participants will be capped at 100.
  Interventions: Diagnostic Test: GeneXpert HBV DNA Viral Load Assay; Diagnostic Test: Dried Blood Spot HBV DNA test

INTERVENTIONS:
Diagnostic Test: GeneXpert HBV DNA Viral Load Assay — The Xpert venous blood HBV DNA viral load assay will be adapted to operate using fingerstick capillary blood samples.
Diagnostic Test: Dried Blood Spot HBV DNA test — HBV DNA viral load will be measured from a fingerstick capillary dried blood spot sample using a gold standard HBV DNA viral load assay

SUMMARY:
This is a cross sectional observational study to asses the performance of two novel HBV DNA testing methodologies; a) dried blood spot sampling and b) fingerstick capillary blood using the Xpert® Hepatitis B Virus viral load assay. Both novel testing methodologies will be compared with venous blood tested using a gold standard HBV DNA assay. The sensitivity and specificity of the two novel testing will be evaluated.

HBV viral load tests are essential to guide antiviral treatment eligibility and effectiveness. However, many people are unable to access these tests, particularly those living in remote or limited resources settings given high cost, or unavailable infrastructure. Simple, affordable and accessible HBV viral load tests are required to increase global access to HBV testing and treatment to meet the WHO HBV elimination targets. The GeneXpert Diagnostic Systems, the most common molecular point-of-care platform globally, has the potential to provide simple and affordable HBV viral load tests. Dried Blood Spot testing is also an affordable and accessible testing methodology particularly suited to remote and resource limited settings. This proof-of-concept study will assess the feasibility and diagnostic performance of Xpert® HBV Viral Load test and Dried Blood Spot testing for the quantitation of HBV DNA from fingerstick capillary samples.

DETAILED DESCRIPTION:
This study will be a cross-sectional observational study and will assess the performance of a novel fingerstick HBV Viral Load and Dried Blood Spot tests within a total of 300 participants who will be recruited across a network of hepatitis clinics in Sydney, Australia. No treatment will be administered as part of this study.

The Xpert HBV cartridge will be adapted to use fingerstick capillary blood instead of processed whole blood, and it's performance measured against a gold standard venous blood HBV DNA assay. Dried Blood Spot HBV DNA testing performance will also be measured against the gold standard venous blood HBV DNA assay.

Secondary objectives of the study are to: 1) evaluate diagnostic performance of the Xpert® HBV Viral Load assay compared to standard of care testing, by patients' hepatitis B e-antigen status (among e-antigen positive and e-antigen negative patients). 2) Evaluate diagnostic performance of the Xpert® HBV Viral Load assay compared to standard of care testing, by HBV treatment status (among treatment naïve patients and those receiving treatment). 3) Evaluate diagnostic performance of the Xpert® HBV Viral Load assay compared to standard of care testing, by HBV DNA levels (among patients with HBV DNA <20 IU/mL; between 20 and 2,000 IU/mL, between 2,000 and 20,000 IU/mL; between 20,000 and 200,000 IU/mL; and >200,000 IU/mL).

ELIGIBILITY:
Inclusion Criteria:

* Have voluntarily signed the informed consent form, 18 years of age or older, HBsAg positive

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from across the network of tertiary hepatitis clinics active in providing HBV clinical care. All participants must meet the inclusion criteria to be eligible to participate in the study.
  Participants will be recruited irrespective of HBV DNA Level, HBeAg or treatment status.
Sampling Method: Non-Probability Sample
Enrollment: 268 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Assess performance of Xpert HBV DNA viral load assay using novel fingerstick capillary blood collection and HBV DNA viral load using fingerstick capillary Dried Blood Spot sample collection. | At completion of enrolment
  Evaluate the diagnostic performance of the Xpert HBV viral load assay and DBS samples using fingerstick capillary blood compared with the gold standard venous blood HBV DNA viral load assay

SECONDARY OUTCOMES:
Evaluate diagnostic performance of the novel tests by hepatitis B e-antigen status | At completion of enrolment
  Evaluate the diagnostic performance of the Xpert HBV viral load assay and DBS samples using fingerstick capillary blood compared with the gold standard venous blood HBV DNA viral load assay by 'Hepatitis B e-antigen status (among e-antigen positive and e-antigen negative patients).
Evaluate diagnostic performance of the novel tests by HBV treatment status | At completion of enrolment
  Evaluate the diagnostic performance of the Xpert HBV viral load assay and DBS samples using fingerstick capillary blood compared with the gold standard venous blood HBV DNA viral load assay by HBV treatment status (among treatment naïve patients and those receiving treatment)
Evaluate diagnostic performance of the novel tests by HBV DNA levels | At completion of enrolment
  Evaluate the diagnostic performance of the Xpert HBV viral load assay and DBS samples using fingerstick capillary blood compared with the gold standard venous blood HBV DNA viral load assay by HBV DNA levels (among patients with HBV DNA <20 IU/mL; between 20 and 2,000 IU/mL, between 2,000 and 20,000 IU/mL; between 20,000 and 200,000 IU/mL; and >200,000 IU/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Gail V Matthews, MBChB, Principal Investigator — The Kirby Institute, University of New South Wales Australia
Locations (6):
- Australia (6):
  - St Vincent's Hospital, Sydney, New South Wales
  - Prince of Wales Hospital, Sydney, New South Wales
  - STORR Liver Centre Westmead Hospital, Sydney, New South Wales
  - Blacktown Hospital, Sydney, New South Wales
  - Liverpool Hospital, Sydney, New South Wales
  - St Vincent's Hospital Melbourne, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No